CLINICAL TRIAL: NCT00170235
Title: Reducing Arm Morbidity Through Physical Therapy Provided Pre- and Post-breast Cancer Surgery
Brief Title: Reducing Arm Morbidity in Pre- and Post-breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Dr Nancy Mayo, McGill University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: SDR-05-017
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Prehabilitation; Rehabilitation; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Prehabilitation (exercises pre surgery)
  Interventions: Other: Prehabilitation
- 2 (Active Comparator): Usual care as provided by the institution
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Prehabilitation — Exercise class pre-surgery
  Arms: 1
Other: Usual care — Exercise booklet, physiotherapy if needed
  Arms: 2

SUMMARY:
The overall aim of this pilot study is to explore the feasibility of a randomized trial to test the effectiveness of physical therapy, provided both pre- and post-surgery, on reducing arm morbidity and increasing health-related quality of life (HRQL) post-surgery.

DETAILED DESCRIPTION:
Breast cancer surgery is one of the most frightening health events a woman can experience. Not only is there fear of cancer and mortality, but also fear of disfigurement and disability arising from the surgery and from the subsequent chemotherapy and radiotherapy. The pre-operative period is a time of great anxiety and in the post-operative period this anxiety is compounded by pain and discomfort associated with the breast and axillary wounds. Lack of knowledge about follow-up treatment leads to fear and anxiety post-surgery. All women experience loss of mobility and function of the arm on the operative side for a period of time ranging from days to months to years. This arm morbidity interferes with participation in usual activities, is an additional source of stress compounding the psychological distress associated with the cancer itself, and has a negative impact on the quality of life.

The post-operative period may not be the most opportune time to introduce interventions to accelerate recovery. Many women will be concerned about perturbing the healing process and may be depressed and anxious as they await extra treatment for the tumor. The pre-operative period may be a more emotionally salient time to intervene in the factors that contribute to recovery.

The process of enhancing functional capacity of the individual to enable him or her to withstand stressors is termed "prehabilitation". This project deals with the effectiveness of prehabilitation with or without post-operative exercise to reduce arm morbidity and increase quality of life following breast cancer surgery.

The overall aim is to explore the feasibility of a randomized trial to test the effectiveness of physical therapy, provided both pre- and post-surgery, on reducing arm morbidity and increasing health-related quality of life (HRQL) post-surgery. The specific objectives of this pilot project are to:

1. estimate recruitment rates for such a trial;
2. estimate compliance to the protocols;
3. pilot the randomization procedures;
4. identify sub-groups of the population with different needs for pre-and post-surgical physical therapy;
5. estimate effect sizes to be used for sample size calculations for the main project and for budget justification.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Diagnosed with breast cancer
* Able to complete questionnaires

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-08; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
participation restriction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mayo, PhD, Principal Investigator — James McGill Professor, Department of Medicine, School of Physical and Occupational Therapy, McGill University
Locations (1):
- Division of Clinical Epidemiology, Montreal, Quebec, Canada

REFERENCES:
- [Background] Mayo NE, Scott SC, Shen N, Hanley J, Goldberg MS, MacDonald N. Waiting time for breast cancer surgery in Quebec. CMAJ. 2001 Apr 17;164(8):1133-8. PMID 11338798
- [Background] Shen N, Mayo NE, Scott SC, Hanley JA, Goldberg MS, Abrahamowicz M, Tamblyn R. Factors associated with pattern of care before surgery for breast cancer in Quebec between 1992 and 1997. Med Care. 2003 Dec;41(12):1353-66. doi: 10.1097/01.MLR.0000100581.88722.6C. PMID 14668668